CLINICAL TRIAL: NCT04353076
Title: Understanding and Managing the Limits of Physiological Tolerance in Heat Vulnerable Canadians During Rest and Physical Exercise
Brief Title: Physiological Responses in Young and Older Adults During a Prolonged Simulated Heatwave
Acronym: HW1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Glen P. Kenny, Full Professor, University Research Chair, University of Ottawa
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: H 05-16-07
Record Dates: First submitted 2020-04-13; First posted 2020-04-20 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Aging; Heat Stress; Physiological Stress
Keywords: Heatwave; Heat-vulnerability; Cooling center; Heat strain; Cardiovascular responses
MeSH Terms: conditions — Heat Stress Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Young adults (Experimental): Young adults exposed to a 9-hour simulated heatwave (40°C, 15% relative humidity)
  Interventions: Other: Simulated heatwave exposure
- Older adults (no cooling) (Experimental): Older adults exposed to a 9-hour simulated heatwave (40°C, 15% relative humidity)
  Interventions: Other: Simulated heatwave exposure
- Older adults (cooling) (Experimental): Older adults exposed to a 9-hour simulated heatwave (40°C, 15% relative humidity) with ambient cooling intervention (i.e., exposure to an air-conditioned room) for hours 5-6.
  Interventions: Other: Simulated heatwave exposure with mid-day cooling

INTERVENTIONS:
Other: Simulated heatwave exposure — Young and older adults (no cooling) are exposed to a 9-hour simulated exposure.
  Arms: Older adults (no cooling); Young adults
Other: Simulated heatwave exposure with mid-day cooling — Older adults (cooling) are exposed to a 9-hour simulated exposure with mid-day ambient cooling.
  Arms: Older adults (cooling)

SUMMARY:
Climate change not only affects the planet's natural resources, but also severely impacts human health. An individual's ability to adequately cope with short- or long-term increases in ambient temperature is critical for maintaining health and wellbeing. Prolonged increases in temperature (heatwaves) pose a serious health risk for older adults, who have a reduced capacity to efficiently regulate body temperature. However, information regarding the impact of age on body temperature regulation during prolonged exposure to extreme heat is lacking, as is research on the effectiveness of interventions aimed at reducing heat strain in such situations. This project will address these important knowledge gaps by exposing healthy young and older adults to a prolonged (9 hour) heat exposure, with conditions representative of heatwaves in temperate continental climates. An additional cohort of older adults will complete the same heatwave simulation but will be briefly (2 hours) exposed to cooler conditions (22-23°C) mid-way through the session (akin to visiting a cooling centre or cooled location). The investigators will evaluate age-related differences in the capacity to dissipate heat via direct air calorimetry (a unique device that permits the precise measurement of the heat dissipated by the human body) and their effect on the regulation of body temperature. The investigators anticipate that older adults will exhibit progressive increases in the heat stored in the body throughout the simulated heatwave, resulting in progressive increases in body core temperature. Further, older adults exposed to brief-mid day cooling will rapidly gain heat upon re-exposure to high ambient temperatures. As a result, by the end of exposure body temperatures will be similar to the group not removed from the heat.

DETAILED DESCRIPTION:
OBJECTIVES Intervention 1: Evaluate the effect of age on whole-body heat storage, body core temperature, and the development of cardiovascular strain and acute inflammation during day-long (9 hours) exposure to simulated heatwave conditions.

Intervention 2: Determine whether short-duration exposure (2 hours) to an air-conditioned environment following extreme heat exposure results in lasting reductions in physiological strain in older adults upon return to the heat.

Hypotheses Intervention 1: Older adults will experience greater heat storage throughout the 9-hour simulated heatwave compared to the younger participants. Consequently, body core temperature will be greater in the older adults and between-group differences will be exacerbated as exposure progresses. We will also explore the secondary hypothesis that differences in body temperature will be paralleled by greater alterations in cardiovascular variables and acute circulatory and intracellular inflammation in the older adults.

Intervention 2: Body heat storage will be exacerbated in the older adults exposed to the cooling centre intervention upon return to the heat (hours 5-6) compared to the older adults from Intervention 1 who remained in the heat. Consequently, body core temperature will be comparable (statistically equivalent) between groups by the end of exposure.

Methods Participants A total of 20 young (age: 18-31 years) and 40 older (age: 64-80 years) adults will be recruited for the proposed project, with an approximately even distribution of men and women in each intervention arm. Young (n = 20) and older (n = 20) adults will complete Intervention 1 and a separate cohort of older adults (n = 20) will complete Intervention 2. Participants will be homogenous for anthropomorphic characteristics as well as habitual physical activity levels as verified via standardized questionnaires.

Experimental Design Pre-trial instructions All participants will be asked to avoid strenuous physical activity and alcohol for 24 hours prior to all preliminary and experimental sessions and to eat a light meal 2 hours before the start of each session. Participants will also be asked to consume a minimum of 500 ml of water the night before and morning of each session to ensure adequate hydration. Adequate hydration will be verified upon arrival to the laboratory (urine specific gravity <1.025). For all sessions, participants will wear athletic shorts (and a sport top for women).

Preliminary screening All participants will complete one preliminary evaluation a minimum of 7 days before the first experimental session. During this session they will be familiarized with all procedures and measurement techniques and will complete the Get Active Questionnaire (GAQ) and the American Heart Association Pre-participation screening Questionnaire to assess their eligibility to participate. The GAQ will also be used to assess habitual activity levels along with the Kohl Physical Activity Questionnaire. Participants will also provide verbal and written informed consent at this time. Body height and mass will be determined via a physician stadiometer and a high-performance weighing terminal, respectively, and from these measurements body surface area will be calculated.

Experimental Protocol (Intervention 1) Each session will commence at 07:00-09:00. Upon arrival to the laboratory, the participant will provide a urine sample for the assessment of urine specific gravity, after which a measurement of nude body mass will be obtained. Participants will then insert a temperature probe for the continuous measurement of rectal temperature. Thereafter, participants will be instrumented for the measurement of skin temperature and 5-lead echocardiogram. Baseline cardiovascular parameters will be evaluated via a brief (~45 min) cardiovascular test battery, performed as follows. Brachial arterial systolic and diastolic pressures reconstructed from arterial pressure waveforms measured at the right middle finger (volume clamp technique) and 5-lead echocardiogram recordings will be collected for 10-min while the participant rests quietly (spontaneous breathing). Immediately thereafter, arterial systolic and diastolic pressures will be measured in triplicate via manual auscultation (~30 sec between measures), after which forearm and calf blood flows on the right side of the body will be measured via automated venous occlusion plethysmography. Throughout the test battery, the participant will be seated with both feet on the floor, except for during the measurements of limb blood flow, where the instrumented limbs will be elevated to facilitate venous drainage. Finally, a venous blood sample and body mass measurement will be obtained.

Participants will then be transferred to the whole-body direct calorimeter chamber, regulated to 40°C and ~10-15% humidity. These conditions were chosen to simulate peak temperatures experienced during heatwaves and are similar to peak conditions in recent heatwaves in North America in 2018 (Ottawa, Ontario; 34°C and 58%, heat index: 41°C) and Europe in 2003 (Paris, France; 38°C and 25%, heat index: 38°C). The participant will rest quietly for 3-hours (hours 1-3) within the calorimeter chamber while whole-body heat production and exchange are measured continuously. At the 3-hour mark, the participant will exit the calorimeter and the brief cardiovascular test battery will be performed again followed by a measurement of body mass. Hours 4-6 will be spent resting in the heat in the thermal chamber adjacent to the calorimeter. During this time, participants will be allowed to consume a light, self-provided lunch with low water content. Tap water will be provided ad libitum via a self-service insulated water cooler located in the thermal chamber. Another cardiovascular battery will then be performed followed by a measurement of body mass. The participant will then re-enter the calorimeter where the final 3 hours will be spent (hours 6-9). At the end of this period, the participants will undergo a fourth and final cardiovascular test battery and a final venous blood sample and body mass measurement will be procured.

Statistical analysis and sample size calculations Primary and secondary variables will be evaluated using linear mixed-effects models. Time will be modelled as a repeated within-subject fixed effect, and age-group will be modelled as a between-subject fixed effect. Pre-heat exposure values of the outcome variable, participant sex, and self-reported weekly physical activity (min/week, as assessed via the GAQ) will be included as covariates. Participant identification will be modeled as a random effect in all analyses. Akaike's information criterion will be used to determine random effect and variance/covariance structures.

Post hoc multiple comparisons will be made on model estimated marginal means. Given the small number of comparisons for each variable, multiplicity corrections will not be employed. Homoscedasticity will be evaluated for all models by visual assessment of residual plots. Approximate normal distribution of residuals will be assessed via visual inspection of histograms and Q-Q plots. Data will be log-transformed in the event that the distribution of residuals meaningfully deviates from normality. For all analyses, alpha will be set at 0.050. Descriptive statistics will be presented as means and standard deviations. Comparisons between groups and/or time-points will be presented as means and 95% confidence intervals [lower limit, upper limit].

An a priori power analysis determined that a total sample size of 19 young and 19 older adults was required to detect a difference in the rate of whole-body heat storage between groups at the end of each calorimeter session (i.e., hours 3 and 9) with 80% statistical power. In lieu of clinically meaningful data (i.e., what would be considered a clinically meaningful change in whole-body heat storage), the standardized effect size (Cohen's d=1.06) was calculated based on the difference in the rate of whole-body heat storage between young and older adults over the final 30-min of a 3-hour heat exposure protocol (young: -2 [26] kJ/hour, older: 43 [54] kJ/hour) in our previous work.

Experimental Protocol (Intervention 2) Experimental design The protocol for Intervention 2 is identical to that of Intervention 1 except that after the first calorimeter session and subsequent cardiovascular battery, participants will exit the thermal chamber and spend ~2 hours (hours 5-6) resting in an air-conditioned room (~23°C, ~50% relative humidity). Similar to Intervention 1, participants will be allowed to eat a small self-provided lunch during this time and consume water (tap) ad libitum. The third cardiovascular battery will also be performed in the cooled environment. As in Intervention 1, participants will then re-enter the calorimeter for the final 3 hours, where they will rest in the heat for the remainder of the experimental session.

Statistical analysis and sample size calculations Statistical analysis for Intervention 2 will be performed to assess whether mid-day exposure to a cooled room results in greater body heat storage following exposure such that physiological responses are similar to those of the non-cooled group by the end of the 9-hour heatwave simulation. Cumulative whole-body heat storage will be evaluated using a linear mixed-effects model with experimental group modelled as a between-subject fixed effect. Cumulative heat storage over the first three hours of the 9-hour exposure will be included as a covariate to account for the influence of any inter- or intra-individual factors (e.g., sex, physical activity levels), measured or unmeasured, impacting whole-body heat exchange and storage. Comparisons of heat storage between groups will be made using model estimated marginal means.

Body core temperature, as estimated by rectal temperature (primary outcome), will be analyzed with a linear mixed effects model with experimental group (two levels: cooling and no-cooling) modelled as a between-subject fixed effect and time as a repeated within-subject fixed effect (0-, 1-, 2-, and 3-hours post-cooling intervention). Like the model for heat storage, rectal temperature at the end of the first calorimetry session (i.e., hour 3 of the 9-hour exposure) will be included as a covariate to account for the influence of any measured or unmeasured inter- or intra-individual factors impacting the body temperature responses to resting heat exposure.

The effect of cooling on rectal temperature will then be assessed via two one-sided tests performed on the mixed-effects model derived estimated marginal means at each timepoint. Equivalence bounds will be set to ±0.3°C, which corresponds to the typical day-to-day variation of core temperature and has been suggested to reflect a meaningful/detectable change in body temperatures in a recent study assessing the influence of cooling strategies on physiological strain in young adults. Secondary variables will be similarly evaluated. The level of significance will be set at P < 0.050. Descriptive statistics will be presented as mean (standard deviation) and comparisons between groups will be presented as mean ± 95% confidence interval.

An a priori power analysis determined that a total sample size of 18 older adults in each group (36 participants total) is required to confirm whether between-group differences in rectal temperature are equivalent within upper and lower bounds of +0.3°C and -0.3°C, respectively, with 80% power. This corresponds to an effect size (Cohen's d) of 1.0, based on the pooled-standard deviation of 0.3°C, determined from published data from our laboratory demonstrating a 0.2°C (SD 0.3) difference in core temperature between young and older adults and a 0.0°C (SD 0.3) difference in core temperature between older adults with and without type 2 diabetes following 3 hours of rest in a hot environment.

ELIGIBILITY:
Inclusion Criteria:

* male or female (non-pregnant) adults with or without a) chronic hypertension (elevated resting blood pressure; as defined by Heart and Stroke Canada and Hypertension Canada), b) type 2 diabetes as defined by Diabetes Canada, with at least 5 years having elapsed since time of diagnosis and or c) obesity as defined by the World Health Organization (Body Mass Index [BMI] greater than or equal to 30).
* non-smoking.

Exclusion Criteria:

* Episode(s) of severe hypoglycemia (requiring the assistance of another person) within the previous year, or inability to sense hypoglycemia (hypoglycemia unawareness).
* Serious complications related to your diabetes (gastroparesis, renal disease, uncontrolled hypertension, severe autonomic neuropathy).
* Uncontrolled hypertension - BP >150 mmHg systolic or >95 mmHg diastolic in a sitting position.
* Restrictions in physical activity due to disease (e.g. intermittent claudication, renal impairment, active proliferative retinopathy, unstable cardiac or pulmonary disease, disabling stroke, severe arthritis, etc.).
* Use of or changes in medication judged by the patient or investigators to make participation in this study inadvisable.
* Cardiac abnormalities identified in your physical health screening form (adults <65 years of age and older; adults <60 years of age and older with diabetes and or hypertension) or during exercise stress testing as assessed by 12-lead (all adults ≥65 years of age and older).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-04-02 (Actual); Study Completion 2021-04-02 (Actual)

PRIMARY OUTCOMES:
Body heat storage | First 3 hours (hours 1-3) of simulated heatwave
  Cumulative amount of heat stored within the body
Body heat storage | Final 3 hours (hours 7-9) of simulated heatwave
  Cumulative amount of heat stored within the body
Rectal temperature | Hour 3 of simulated heatwave
  Index of core body temperature
Rectal temperature | Hour 9 of simulated heatwave
  Index of core body temperature

SECONDARY OUTCOMES:
Heart rate | Hour 3 of simulated heatwave
  Measured continuously throughout exposure
Heart rate | Hour 9 of simulated heatwave
  Measured continuously throughout exposure
Systolic blood pressure | Hour 3 of simulated heatwave
  Arterial blood pressures measured via manual auscultation
Systolic blood pressure | Hour 9 of simulated heatwave
  Arterial blood pressures measured via manual auscultation
Diastolic blood pressure | Hour 3 of simulated heatwave
  Arterial blood pressures measured via manual auscultation
Diastolic blood pressure | Hour 9 of simulated heatwave
  Arterial blood pressures measured via manual auscultation
Mean arterial pressure | Hour 3 of simulated heatwave
  calculated as 1/3 * systolic blood pressure + 2/3 diastolic blood pressure
Mean arterial pressure | Hour 9 of simulated heatwave
  calculated as 1/3 * systolic blood pressure + 2/3 diastolic blood pressure
Rate pressure product | Hour 3 of simulated heatwave
  Calculated as systolic blood pressure * heart rate
Rate pressure product | Hour 9 of simulated heatwave
  Calculated as systolic blood pressure * heart rate
Cardiac baroreflex sensitivity | Hour 3 of simulated heatwave
  Determined from beat-to-beat arterial pressures and heart rate (volume-clamp technique)
Cardiac baroreflex sensitivity | Hour 9 of simulated heatwave
  Determined from beat-to-beat arterial pressures and heart rate (volume-clamp technique)
Change in plasma volume | Hour 9 of simulated heatwave
  Determined from venous blood samples
Heart rate variability: SDNN | Hour 3 of simulated heatwave
  Standard deviation of successive normal R-R intervals
Heart rate variability: SDNN | Hour 9 of simulated heatwave
  Standard deviation of successive normal R-R intervals
Heart rate variability: RMSSD | Hour 3 of simulated heatwave
  Root mean squared standard deviation of successive normal R-R intervals
Heart rate variability: RMSSD | Hour 9 of simulated heatwave
  Root mean squared standard deviation of successive normal R-R intervals
Circulating inflammatory and stress markers | Hour 9 of simulated heatwave
  Tumor necrosis factor alpha, Interleukin 6, C-reactive protein
Intracellular inflammatory and stress markers | Hour 9 of simulated heatwave
  Tumor necrosis factor alpha, Interleukin 6, Heat shock proteins 70 and 90

CONTACTS AND LOCATIONS:
Overall Officials: Glen P Kenny, PhD, Principal Investigator — University of Ottawa; Ronald J Sigal, MD, MPH, Principal Investigator — University of Calgary
Locations (1):
- University of Ottawa, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Journeay WS, McCormick JJ, King KE, Garrett JM, O'Connor FK, Hutchins KP, Meade RD, Kenny GP. Serum endothelial monocyte-activating polypeptide-II response after 9 h of passive heat exposure: influence of age, diabetes, or hypertension. Am J Physiol Regul Integr Comp Physiol. 2026 Feb 1;330(2):R119-R125. doi: 10.1152/ajpregu.00307.2025. Epub 2026 Jan 9. PMID 41512819
- [Derived] Garrett JM, McCormick JJ, King KE, Meade RD, Boulay P, Sigal RJ, O'Connor FK, Kenny GP. Irisin and betatrophin responses to 9 h of passive heat exposure: Influence of age, hypertension, and type 2 diabetes. Physiol Rep. 2025 Jun;13(12):e70411. doi: 10.14814/phy2.70411. PMID 40554659
- [Derived] Lee B, Meade R, Davey S, Thake C, McCormick J, King K, Kenny GP. Effect of brief ambient cooling on serum stress biomarkers in older adults during a daylong heat exposure: a laboratory-based heat wave simulation. Appl Physiol Nutr Metab. 2025 Jan 1;50:1-8. doi: 10.1139/apnm-2024-0476. PMID 40036754

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-11): https://cdn.clinicaltrials.gov/large-docs/76/NCT04353076/Prot_SAP_001.pdf